CLINICAL TRIAL: NCT06862700
Title: Association Between Vasopressor Exposure Levels and 30-Day Mortality in Patients Receiving ECMO Support for Cardiogenic Shock: A Prospective Multicenter Cohort Study
Brief Title: Effect of Reduced Vasopressors on Mortality in ECMO-supported Cardiogenic Shock Patients
Acronym: VREM-CS
Status: Recruiting | Type: Observational
Sponsor: Xiaotong Hou (Other)
Responsible Party: Sponsor-Investigator, Xiaotong Hou, Clinical professor, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Other Study IDs: 2025038x
Record Dates: First submitted 2025-02-26; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Cardiogenic Shock; Extracorporeal Membrane Oxygenation; Vasopressors; Hemodynamic Management; Critical Care; Heart Failure
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High VIS Group: High VIS Group: Patients with an average Vasoactive-Inotropic Score (VIS) >10 from 12 hours post-ECMO initiation to weaning.
  Interventions: Other: Vasopressor Exposure Levels
- Low VIS Group: Low VIS Group: Patients with an average Vasoactive-Inotropic Score (VIS) ≤10 from 12 hours post-ECMO initiation to weaning.
  Interventions: Other: Vasopressor Exposure Levels

INTERVENTIONS:
Other: Vasopressor Exposure Levels — This is an observational study with no active intervention. The study evaluates the association between natural variations in vasopressor exposure levels (measured by Vasoactive-Inotropic Score, VIS) and clinical outcomes in patients receiving VA-ECMO for cardiogenic shock.
  Other Names: Vasoactive-Inotropic Score (VIS)

SUMMARY:
The goal of this observational study is to learn about the association between vasopressor exposure levels and outcomes in adults with cardiogenic shock receiving VA-ECMO. The main question it aims to answer is:

Does reduced exposure to vasopressors lower the 30-day mortality in patients with cardiogenic shock when receiving ECMO support? Participants who are receiving ECMO support for cardiogenic shock as part of their regular medical care will have their data collected, including information about their vasopressor use and mortality outcomes, over the course of the study.

DETAILED DESCRIPTION:
The study will enroll 534 patients from multiple centers who require VA-ECMO for cardiogenic shock. Patients will be stratified into two groups based on their average Vasoactive-Inotropic Score (VIS) from 12 hours post-ECMO initiation to weaning: a high-dose group (VIS >10) and a low-dose group (VIS ≤10). The primary outcome is 30-day all-cause mortality. Secondary outcomes include hospital survival rate, duration of mechanical ventilation, ICU and hospital length of stay, and ECMO-related complications. Hemodynamic parameters and laboratory biomarkers will be monitored. The study aims to identify optimal hemodynamic management strategies, including ECMO flow rates, blood pressure targets, and vasopressor dosing, to improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with cardiogenic shock requiring VA-ECMO support.
* First-time ECMO initiation.
* Venoarterial ECMO (VA-ECMO) as the initial mode.

Exclusion Criteria:

* Age <18 years.
* Severe pulmonary hypertension.
* Vasopressor use for non-shock indications (e.g., bleeding, post-cardiopulmonary bypass vasoplegia).
* Severe missing data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At participating centers, adult patients with cardiogenic shock require venoarterial extracorporeal membrane oxygenation (VA-ECMO) support, meeting specific hemodynamic and end-organ dysfunction criteria.
Sampling Method: Non-Probability Sample
Enrollment: 534 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
30-Day All-Cause Mortality | From ECMO initiation through hospital discharge (assessed up to 6 months).
  The proportion of patients who die from any cause within 30 days following ECMO initiation.

SECONDARY OUTCOMES:
In-Hospital Survival Rate | From ECMO initiation through hospital discharge (assessed up to 6 months).
  The proportion of patients who survive to hospital discharge.
ECMO-Related Complications | From ECMO initiation through hospital discharge (assessed up to 6 months).
  The incidence of ECMO-related complications, including bleeding, thrombosis, infection, and mechanical failures.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Du, MD, Study Chair — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No